CLINICAL TRIAL: NCT06382922
Title: Prospective, Observational Study of the Role of Primary Antifungal Prophylaxis to Prevent Invasive Aspergillosis in Elderly Patients With Acute Myeloid Leukemia Undergoing Consolidation Therapy
Brief Title: Role of Antifungal Prophylaxis in Elderly Patients With Acute Myeloid Leukemia During Consolidation Therapy
Status: Recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Maria Ilaria Del Principe, Associate Professor, University of Rome Tor Vergata
Other Study IDs: PAPAML022019
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Invasive Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In previous retrospective study (SEIFEM 2016 study) the investigators evaluated the incidence of proven/probable invasive aspergillosis (IA) and the role of mold active primary antifungal prophylaxis (PAP) in a "real life" setting of acute myeloid leukemia (AML )patients receiving intensive consolidation therapy. All cases of proven/probable IA, observed during consolidation chemotherapy in adult and pediatric AML patients between 2011 and 2015, were retrospectively collected in a multicenter study involving 38 Italian hematologic centers. The investigators observed 56 (2.2%) cases of IA [43 probable (1.7%) and 13 proven (0.5%)]. The overall mortality rate and the mortality rate attributable to IA (AMR) on day 120 were 16% and 9%, respectively. In multivariate analysis, parameters that influenced the outcome were age ≥60 years and treatment with high doses of cytarabine (HDAC).

The investigators also observed that centers involved in this survey had different antifungal policies during the AML consolidation phase. The results from this study show that in a large real-world setting the mold active PAP, with itraconazole or posaconazole, decreases the rate of IA after consolidation course.

In SEIFEM 2016 study the investigators demonstrated that the incidence of IA during the AML consolidation is low. However, the mortality is not negligible, mainly in older patients. Further, a sub-analysis in the subset of patients older than 60 years demonstrated that patients who didn't receive mold active prophylaxis had higher incidence of IA than patients who received mold active prophylaxis (15% vs 6%). Therefore, as prophylaxis seems to prevent IA in consolidation, further studies should be performed especially in elderly patients treated with HDAC to confirm our data and to identify the subset of patients who require PAP.

DETAILED DESCRIPTION:
Evaluate the protective role of mold active PAP in patients older than 60 years underwent to chemotherapy of consolidation with intermediate or high doses of cytarabine

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national/local laws
* Patients aged older than 60 years underwent to consolidation course with intermediate/high doses of cytarabine

Exclusion Criteria:

• Diagnosis of IA during induction course and previous antifungal treatment

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Considering our previous results and that in the subset of patients older than 60 years patients, who didn't receive mold active prophylaxis had higher incidence of IA than patients who received mold active prophylaxis (15% vs 6%), we calculated that sample side should be 300 patients for arms. This sample size achieves 90% power to detect a difference of 10% .
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of proven, probable and possible IA in patients enrolled in the study in both groups of patients | 60 months
  rate of IA

SECONDARY OUTCOMES:
overall mortality rate | 60 months
  rate

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ilaria Del Principe, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- Tor Vergata University, Roma, RM, Italy